CLINICAL TRIAL: NCT03550885
Title: Diet Modulation of Bacterial Sulfur and Bile Acid Metabolism and Colon Cancer Risk
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Rush University Medical Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lisa Tussing-Humphreys, Assistant Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2016-0495; 1R01CA204808-01 (NIH)
Record Dates: First submitted 2018-05-24; First posted 2018-06-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: microbiome, human; bile acids and salts; diet, western
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Taurine

STUDY DESIGN:
Intervention Model Description: The proposed study will utilize a randomized, crossover, controlled feeding trial design composed of two experimental diets: (1) animal-based, high in taurine and saturated fat (HT-HSAT) and (2) plant-based, low in both taurine and saturated fat (LT-LSAT) (each consumed for 21 days with a minimum 3-week washout between diets).
  At baseline and post-diet (day 22) for each of the two 3-week diets, subjects will undergo a flexible sigmoidoscopy, fasting and non-fasting blood draw, and provide a stool sample.
Who Masked: Investigator
Masking Description: All study personnel, excluding those directly involved with meal preparation, will be blinded to the subjects' diet sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High taurine and saturated fat diet (Experimental): This is a 3-week controlled isocaloric diet containing approximately 125 mg taurine, 40% of calories from fat, 15% of calories from saturated fat, 25% of calories from protein (4:1 animal to plant grams of protein), and 11.5 grams fiber/1000 calories.
  Interventions: Other: High taurine and saturated fat diet
- Low in taurine and saturated fat diet (Experimental): This is a 3-week controlled isocaloric diet containing approximately 7 mg taurine, 36% of calories from fat, 8% of calories from saturated fat, 13% of calories from protein (3:1 plant to animal grams of protein), and 13.5 grams fiber/1000 calories.
  Interventions: Other: Low in taurine and saturated fat diet

INTERVENTIONS:
Other: High taurine and saturated fat diet — This is a 3-week (21 day) isocaloric Western-type diet with all meals, snacks, beverages and condiments provided.
  Arms: High taurine and saturated fat diet
Other: Low in taurine and saturated fat diet — This is a 3-week (21 day) isocaloric largely plant-based diet with all meals, snacks, beverages and condiments provided.
  Arms: Low in taurine and saturated fat diet

SUMMARY:
Determine in the context of a controlled crossover diet-intervention trial the role of taurocholic acid metabolism by gut bacteria in African American subjects at elevated risk for colorectal cancer (CRC). Two isocaloric diets, an animal-based diet high in taurine and saturated fat (HT-HSAT) and a plant-based, low in taurine and low saturated fat (LT-LSAT) will be used to determine the extent to which the relationship between diet (independent variable) and mucosal markers of CRC risk including epithelial proliferation, oxidative stress, DNA damage, and primary and secondary bile acid pools and biomarkers of inflammation (dependent variables) is explained by the abundance of sulfidogenic bacteria and hydrogen sulfide (H2S) concentrations &/or deoxycholic acid (DCA) and DCA-producing bacteria clostridium scindens (mediator variables).

DETAILED DESCRIPTION:
Our research is designed to determine mechanistically why consumption of a high red meat and saturated fat diet imparts risk for CRC development and to demonstrate that primary microbial risk factors (sulfidogenic and bile acid metabolizing bacteria) are modifiable by diet. The focus is on taurine, an overlooked sulfur amino acid (SAA) that is abundant in red meat or provided by bacterial deconjugation of the bile salt TCA, which is increased in subjects consuming a diet high in saturated fat. Rationale for focusing the diet intervention study on AAs comes from the previously mentioned observation that a taurine respiring bacterium distinguished AA but not NHW CRC patients from healthy controls, and the previous work by PI Gaskins in AA subjects focused on mechanisms underlying the increased risk for CRC associated with consumption of a Western type diet.

Our strong collection of past publications and new preliminary data support our hypothesis that dietary sources of organic sulfur increase the abundance of microbes that generate H2S through taurine metabolism and that H2S activates proinflammatory pathways and serves as a genotoxin in the colonic mucosa. We're examining, for the first time bacteria that utilize taurine, which can be provided directly from red meat or indirectly through TCA in response to saturated fat. Our study will be the first to examine the consequences of such specific dietary manipulation on genotoxic or inflammatory pathways implicated in CRC development in at-risk AAs.

Our results will provide novel information regarding the in vivo interactions between diet and cancer that heretofore have not been explored in humans, particularly AAs. Food taurine content is not currently provided in either the University of Minnesota Nutrition Data System for Research (NDSR) or the USDA Standard Reference (USDA SR) nutrient databases, which are the gold standard sources for the nutrient content of food. Evidence that taurine is capable of inducing biomarkers of CRC risk through promoting growth of Sulfidogenic B. wadsworthia or other untargeted bacteria would be an important novel observation justifying the addition of this SAA to these nutrient databases. If our hypothesis is substantiated, simple vigilance of taurine intake might diminish susceptibility to CRC in all individuals, especially AAs at elevated risk. Further, if our hypothesis is upheld, it might be possible to reduce risk not only by dietary intervention but also by microbiota modification (potentially through pre-, pro- or synbiotics). Finally, if our study reveals particular modes of bacterial sulfur or bile acid metabolism correlating with epithelial proliferation or inflammation in AAs, the endpoints identified can potentially predict non-invasively elevated risk individuals who should be: a) advised on specific dietary interventions (those investigated herein); b) offered specific therapy to reduce risk; or c) counseled on regular colonoscopic screening

ELIGIBILITY:
Inclusion Criteria:

1. Adult African American;
2. Obese (defined as BMI 30 - < 50 kg/m2);
3. Age between 45 - 75 years old;
4. Patients with an increased risk for CRC, defined as 3 or more adenomatous polyps or adenomatous polyp > 1cm within 5-yrs of enrollment;
5. An elevated C-reactive protein (CRP) (defined as > 3 mg/l)
6. Participants must be in good general health, not expecting major lifestyle changes in the next 6 months and willing to maintain their current activity level throughout the duration of the study.
7. Women only: Post-menopausal (natural or surgical) defined as no menstruation in the past 6 months

Exclusion Criteria:

1. BMI < 30 or > 50 kg/m2 (for those interested and eligible, verify BMI by measuring weight and height, complete the screening consent form before assessing these measures)
2. Weight > 450 lbs. (max weight for the body composition scanner)
3. Race other than African American
4. Women only: at least one menstrual period in the past 6 months
5. Current malignancy except non-melanoma skin cancer that has been removed
6. Current gastrointestinal (GI) illness other than gastroesophageal reflux disease or hemorrhoids (such as celiac disease, inflammatory bowel disease, malabsorptive bariatric procedures, etc.)
7. Chronic liver or kidney disease (elevated liver tests >3 times normal or creatinine above 2.0 mg/dl)
8. History of cardiac disease (such as admission for congestive heart failure within the past 5 years, or being on anticoagulants for heart disease, or having an ejection fraction <25%, etc.)
9. Positive genetic test for inherited polyposis syndromes (such as familial adenomatous polyps, hereditary non-polyposis colon cancer syndromes, etc)
10. Alcoholism or illicit drug use
11. Antibiotic use within the past 2 months
12. Regularly taking medications that may interfere with normal digestion (such as acarbose, cholestyramine, Orlistat, aspirin doses that exceed 81mg/day or 325 mg every other day)
13. Anticoagulant use or other factors that increase endoscopic risks
14. Non-English speaking
15. Pregnant or breast feeding
16. Dietary supplement use including pre- or probiotics within the past month
17. History of intestinal cancer, inflammatory bowel disease, celiac disease, or malabsorptive bariatric surgery
18. Inflammatory or connective tissue diseases (such as lupus, scleroderma, rheumatoid arthritis, etc.)

21. Prior perforation at colonoscopy or gastrointestinal bleeding due to biopsies of the colon 22. Therapeutic or vegetarian diet 23. Food allergy/aversions to any foods in included in the trial 24. Any medical condition, which, in the opinion of the investigator, could adversely affect the subject's participation in the trial, or affect the trial integrity

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in the mucosal abundance of bacterial genes associated with sulfur and bile acid metabolism | Baseline and post-diet (day 22) for each of the two 3-week diets
  Mucosal abundance of bacterial genes associated with sulfur and bile acid metabolism will be measured by quantitative polymerase chain reaction of 16S rRNA and functional genes with biopsy DNA.

SECONDARY OUTCOMES:
Change in bile acid metabolism | Baseline and post-diet (day 22) for each of the two 3-week diets
  Bile salt hydrolase and bile acid 7a-dehydroxylating activities will be measured in stool samples
Change in serum bile acids | Baseline and post-diet (day 22) for each of the two 3-week diets
  Measurement of serum bile acids using electrospray-ionization mass spectrometry to indicate the extent of taurine-conjugation of bile acids, ratio of conjugated: unconjugated bile acids and levels of secondary bile acids absorbed from the gut
Change in colonic mucosal inflammation | Baseline and post-diet (day 22) for each of the two 3-week diets
  Gene expression of tumor-necrosis factor-alpha, Interleukin-6, and Cox-2
Change in DNA damage | Baseline and post-diet (day 22) for each of the two 3-week diets
  By COMET fluorescence hybridization assay together with in situ staining for 8-oxo-7,8-dihydro-2'-deoxyguanosine (8-oxodG), an oxidative DNA lesion, and the expression of its repair enzyme 8-oxoguanine DNA-glycosylase (OGG1; ab91421), XRCC1 [33-2-5] ab1838), which coordinates the action of DNA ligase III, polymerase beta, and poly-ADP-ribose polymerase in the BER pathway and the apurinic/apyrimidinic endonuclease Ape1 (ab2717), a multifunctional protein that protects cells from oxidative stress via its DNA repair, redox, and transcription regulatory activities
Change in colonocyte proliferation | Baseline and post-diet (day 22) for each of the two 3-week diets
  Immunohistochemistry, Ki-67

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Tussing-Humphreys, PhD, MS, RD, Principal Investigator — University of Illinois at Chicago; Ece Mutlu, MD, MS, MBA, Principal Investigator — Rush University Medical Center; H. Rex Gaskins, PhD, Principal Investigator — University of Illinois at Urbana-Champaign; Jason Ridlon, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Rush University Medical Center and University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form: Rush Aim 2 Consent (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03550885/ICF_002.pdf
  • Informed Consent Form: UIC Aim 2 Consent (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT03550885/ICF_003.pdf